CLINICAL TRIAL: NCT02042807
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled Study to Investigate the Efficacy and Safety of MCS® in Prostate Cancer Prevention
Brief Title: To Evaluate the Effect of MCS® in Prostate Cancer Prevention
Acronym: MCS-8
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Health Ever Bio-Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MCS-8-II-TWN
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Placebo (Placebo Comparator): placebo arm
  Interventions: Drug: Placebo
- MCS® 15 mg/day (Active Comparator): MCS® soft capsule
  Interventions: Drug: MCS®
- MCS® 30 mg/day (Active Comparator): MCS® soft capsule
  Interventions: Drug: MCS®

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: MCS®
  Arms: MCS® 15 mg/day; MCS® 30 mg/day

SUMMARY:
To evaluate the effect of MCS® compared with placebo in reducing the risk of biopsy-detectable prostate cancer in high-risk subjects after 104 weeks (24 months) of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. high-risk subjects of prostate cancer.
2. Male subject with age from 50 to 75 years old.
3. Subject is able to understand and willing to comply with the study procedures and has signed the informed consent form (ICF).

Exclusion Criteria:

1. Subjects who are or will be taking long-term hormonal agents that may affect the normal physiology of sex hormone function.
2. Subjects with a PSA > 10.0 ng/ml.
3. Subjects with a history of prostate cancer.
4. Subject participated in another investigational agent study in the past 30 days or is planning to do so during the study period.
5. Subjects are considered ineligible for the study as judged by the investigator.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Estimated)
Dates: Start 2014-10; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative biopsy-detectable prostate cancer rate | Week 104 (Month 24)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, National Taiwan University Hospital, Taipei, Taiwan